CLINICAL TRIAL: NCT02098902
Title: Randomized Controlled Trial of a Sugar-Sweetened Beverage Intervention in Overweight Mothers and Their Children Ages 3-5
Brief Title: Trial of a Sugar-Sweetened Beverage Intervention in Overweight Mothers and Their Children Ages 3-5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-0547
Record Dates: First submitted 2014-03-25; First posted 2014-03-28 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obesity; Overnutrition; Weight Loss; Body Weight; Nutrition Disorders
MeSH Terms: conditions — Overweight; Obesity; Overnutrition; Weight Loss; Body Weight; Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smart Moms Intervention (Experimental): This arm will receive the Smart Moms intervention immediately following randomization.
  Interventions: Behavioral: Smart Moms Intervention
- Waitlist control group (No Intervention): This arm will receive a modified version of the Smart Moms intervention after the 6-month assessment.

INTERVENTIONS:
Behavioral: Smart Moms Intervention — Reduction in child sugar-sweetened beverage consumption and maternal caloric beverage consumption, in addition to self-selected 100-calorie dietary and physical activity changes made by the mother to promote modest weight loss. Content will be delivered via one in-person group meeting, weekly online lessons, and weekly text messages. Mothers will self-monitor their weight and their own and their child's beverage consumption via text message every 2-3 days.
  Arms: Smart Moms Intervention

SUMMARY:
The purpose of this study is to test the effect of a novel six-month behavioral program to reduce sugar-sweetened beverage consumption among preschoolers and their mothers. The behavioral intervention tested will be delivered via a mobile-based website, text messages and email in addition to one face-to-face group meeting. The intervention will be compared to a waitlist control group. Participants will be 42 overweight/obese mothers and their children ages 3-5 living in the Chapel Hill/Raleigh/Durham area. Sugar-sweetened beverage consumption and weight in both children and mothers will be measured at three- and six-months post-randomization. It is hypothesized that children randomized to the intervention will have a greater reduction in sugar-sweetened beverage consumption at 6 months compared to children randomized to the control group.

DETAILED DESCRIPTION:
Obesity in young children remains a significant public health issue. Interventions targeting this age group are needed, but few have been successful. The most effective childhood obesity prevention interventions for young children thus far have involved significant parent engagement, suggesting that family-based interventions that take into account the needs of both parents and children are needed. But, 2 out of 3 adults are either overweight or obese, and the risk of obesity increases with at least one child under the age of 5 in the home. So not only is obesity among adults high, but maternal obesity is one of the strongest predictors of child obesity, meaning that intervening with overweight and obese mothers could be an effective way of preventing the development of obesity in their young children.

Many family-based or parent-targeted interventions conducted thus far have broadly targeted dietary intake and physical activity, but only a handful have had success in changing child behavior. Interestingly, when evaluating the dietary determinants of childhood obesity, sugar-sweetened beverage (SSB) consumption is most consistently associated with obesity across studies, more so than overall caloric intake, fruit and vegetable consumption, and intake of added dietary fats. Consumption of SSBs makes up 5-18% of preschoolers' recommended daily energy intake, with an average of 176 calories a day consumed from drinks such as caloric carbonated beverages, fruit drinks, sport drinks, and 100% fruit juice. Few interventions have targeted a reduction in SSBs and fruit juice in children, but results from a study in children ages 4-12 found that replacing SSBs with noncaloric beverages can lead to a lower increase in BMI z-scores over time. Reducing SSB consumption in adults is equally as important as in children, because adults consume 21% of their calories from SSBs alone, and consumption of SSBs is associated with a higher risk of obesity, non-alcoholic fatty liver disease, diabetes, the metabolic syndrome, and cardiovascular disease. Several adult intervention studies have shown that replacing caloric beverages, including SSBs, with water or noncaloric beverages can lead to weight loss in the absence of other prescribed changes.

While the research indicates that reducing SSB consumption in children and adults can lead to changes in weight, what is not yet known is if a mother-targeted behavioral intervention can successfully reduce intake of SSBs and fruit juice in preschool-aged children. Because mothers face many barriers to weight control behavior change, including time demands and lack of childcare, there is a need for interventions that are uniquely targeted to the needs of mothers and children, such that they minimize mothers' need to travel, prevent them from having to rearrange their schedules, and minimize the amount of time spent in participation in order to be successful at weight loss and changing their own and their child's behaviors.

This intervention has been developed to focus on changing a small set of behaviors, primarily SSB consumption, in mothers and their children ages 3-5. Guided by Social Cognitive Theory, the intervention will target increases in self-efficacy, outcome expectations, limit setting, and self-monitoring, and decreases in perceived barriers to behavior change. In addition, mothers will be asked to make other small changes in her own behavior to promote modest weight losses. The evidence from traditional behavioral weight loss intervention research has been adapted to focus on making small diet and physical activity changes more suitable for mothers of young children and to be delivered primarily via a mobile-based website and text messaging to reduce time demands and increase adherence. Mother-child dyads (N=42) will be randomized to either the Smart Moms intervention group (n=21) or to a waitlist control group (n=21) that will receive a modified version of the intervention after the 6-month assessment.

ELIGIBILITY:
Inclusion Criteria:

* The parent is female
* The mother has a BMI between 25 and 50
* The mother has a smartphone with data and text messaging plan
* The child is between the ages of 3-5
* The child consumes at least 12 ounces of sugar-sweetened beverages/100% fruit juice per day

Exclusion Criteria:

* The mother cannot speak or read English
* They cannot participate in assessment visits at the UNC Weight Research Program
* The mother is currently participating in another weight loss program
* The mother is pregnant or planning to become pregnant in next 6 months
* They are planning on moving out of the study area in the next 6 months
* The mother has a diagnosis of schizophrenia or bipolar disorder, or hospitalization for a psychiatric diagnosis in the past year
* The mother has excessive intake of alcoholic beverages defined as >14 servings per week or they report a diagnosis of substance or alcohol abuse (on screening survey)
* The mother is unable to safely participate in alternatives to sedentary behavior including standing and walking

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in child sugar-sweetened beverage consumption from baseline to 6 months | Baseline, 6 months
  The primary outcome is the child's average ounces per day of sugar-sweetened beverage consumption change from baseline to 6 months. Sugar-sweetened beverage consumption includes all beverages sweetened with sugar in addition to 100% fruit juice. It will be measured using a 24-hour dietary recall during the in-person assessment visit. A staff member trained to conduct dietary recalls will conduct a mother-reported dietary recall for the child. Dietary data will be entered into the Nutrition Data System for Research (NDSR), which will produce a report that includes intake of sugar-sweetened beverages in ounces per day.

SECONDARY OUTCOMES:
Change in maternal caloric beverage consumption from baseline to 3 months | Baseline, 3 months
  A secondary outcome is the mother's average ounces per day of caloric beverage consumption change from baseline to 3 months. Caloric beverage consumption includes sugar-sweetened beverages, fruit juices, and alcoholic drinks. It will be measured using a 24-hour dietary recall during the in-person assessment visit. A staff member trained to conduct dietary recalls will conduct a dietary recall with the mother. Dietary data will be entered into NDSR, which will produce a report that includes intake of caloric beverages in ounces per day.
Change in maternal weight from baseline to 6 months | Baseline, 6 months
  Mothers will be weighed wearing shorts and without shoes using a calibrated digital Tanita scale. Trained study staff will conduct these measurements following a standardized protocol. Two measures will be completed and the average of the two will be used. Percent weight loss from baseline to 6 months will be calculated and used as the secondary outcome measure.

OTHER OUTCOMES:
Change in child BMI z-score from baseline to 6 months | Baseline, 6 months
  Change in child BMI z-score from baseline to 6 months will also be evaluated in this study. Children will be weighed wearing shorts and without shoes using a calibrated digital Tanita scale. Children's height will be measured at each time point using a wall-mounted stadiometer. Trained study staff will conduct these measurements following a standardized protocol. BMI z-score will be calculated using a program developed by the Centers for Disease Control (CDC).

CONTACTS AND LOCATIONS:
Overall Officials: Brooke T Nezami, MA, Principal Investigator — University of North Carolina, Chapel Hill; Deborah F Tate, PhD, Study Director — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Nezami BT, Lytle LA, Tate DF. A randomized trial to reduce sugar-sweetened beverage and juice intake in preschool-aged children: description of the Smart Moms intervention trial. BMC Public Health. 2016 Aug 19;16(1):837. doi: 10.1186/s12889-016-3533-8. PMID 27542357